CLINICAL TRIAL: NCT03010800
Title: Randomized, Crossover Feasibility Study of a Device to Prevent Female Urinary Stress Incontinence
Brief Title: A Feasibility Device Study to Prevent Female Urinary Stress Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Watkins Conti Products. Inc. (Industry)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WCP001
Record Dates: First submitted 2016-12-27; First posted 2017-01-05 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-06

CONDITIONS: Stress Incontinence, Female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Yoni.Fit (Experimental): Subjects will perform the Abbreviated Pad Test with the Yoni.Fit first, then without the Yoni.Fit.
  Interventions: Device: With Yoni.Fit
- Without Yoni.Fit (Experimental): Subjects will perform the Abbreviated Pad Test without the Yoni.Fit first, then with the Yoni.Fit.
  Interventions: Device: Without Yoni.Fit

INTERVENTIONS:
Device: With Yoni.Fit — Abbreviated Pad Test with Yoni.Fit first, then without Yoni.Fit.
  Arms: With Yoni.Fit
Device: Without Yoni.Fit — Abbreviated Pad Test without Yoni.Fit, then with Yoni.Fit.
  Arms: Without Yoni.Fit

SUMMARY:
This study will test the acute efficacy of an investigational device (Yoni.Fit) in a clinical trial of women with incontinence in a standardized set of challenges performed with and without the device in place.

DETAILED DESCRIPTION:
1. Potential subjects will be pre-qualified by a 6-item questionnaire, the validated Questionnaire for Urinary Incontinence Diagnosis (QUID). This questionnaire has 3 questions each referring to the seriousness of Stress Urinary Incontinence (SUI) and of Urge Urinary Incontinence (UUI). Subjects will be accepted if their SUI score is 5 or greater and is greater than the UUI score. For privacy reasons, these scores will not be retained. Subjects will then be given an appointment. Subjects will be instructed to wear comfortable athletic type wear and not to drink any fluid for two hours prior to their appointment.
2. When subjects appear for their appointment, subjects will be administered the informed consent by the Study Coordinator. All paperwork will be pre-numbered with a code that will link to the subject name. The key will be kept confidential by the Study Coordinator. They will be instructed to empty their bladders and will be given a liter of water or other drink and instructed to drink it over a 15-20 minute time period. An abbreviated patient history will be obtained for the purpose of establishing whether the subject meets the inclusion criteria and is not disqualified by meeting the exclusion criteria. The subject will again fill out the QUID questionnaire. The inclusion criteria are a SUI score of 5 or greater, predominately SUI (SUI score>UUI score) and age between 25 and 65. Exclusion criteria are predominantly UUI, prolapse greater than mild, hysterectomy or other pelvic floor surgery other than a Caesarian section, diabetes, pregnant, BMI>35 or unable to perform ten "jumping jack" exercises. Patients will be administered three additional questionnaires in order to compute a Severity Score. These questionnaires are the Urinary Distress Inventory (UDI), Urinary Impact Questionnaire (UIQ) and the Incontinence Severity Index (ISI). The scores will be multiplied together to provide the Severity Score.
3. Patients will be randomized to Group A or Group B to participate in an abbreviated Pad Test. Group A will perform the test with the Yoni.Fit device in place then repeat the test without the device. Group B will perform the test without the Yoni.Fit device in place then repeat the test with the device in place. This test has been validated (5). An hour after finishing the liter of liquid, the subject is given a tared incontinence pad, which is then put in place. She then engages in the following mild exercise challenges..

   1. Stand from sitting 10 times.
   2. Cough vigorously while standing.
   3. Bend down to pick up small object.
   4. Perform ten jumping jacks. The subject then will remove pad, place into bag and seal. The Experimenter will then weigh pad. The subjects will be randomized so that half will perform the Abbreviated Pad Test with the Yoni.Fit device in place followed by repeating without the device in place. The other half will perform the challenges in the reverse order.
4. The experimenter will calculate a change in score, which is the weight of the pad worn without the device in place minus the tare weight of the pad divided by the weight of the pad with the device in place minus the tare weight of the pad. In case no urine is released with the device in place, the Improvement Score will be defined as "1000". A Release Change will also be calculated as the net weight without the device in place minus the weight with the device in place divided by the net weight released without the device in place.

ELIGIBILITY:
Inclusion Criteria:

* Urinary Incontinence Diagnosis (QUID). This questionnaire has 3 questions each referring to the seriousness of Stress Urinary Incontinence (SUI) and of Urge Urinary Incontinence (UUI). Subjects will be accepted if their SUI score is 5 or greater and is greater than the UUI score.

Exclusion Criteria:

* Refusal to sign the informed consent document
* SUI score is less than 5 or is less than the UUI score.
* Predominantly UUI
* Prolapse greater than mild
* Hysterectomy or other pelvic floor surgery other than a Caesarian section
* Diabetes,
* Pregnant,
* BMI>35 or unable to perform ten "jumping jack" exercises.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang W, Wang T, Zong H, Zhang Y. Efficacy and Safety of Tension-Free Vaginal Tape-Secur Mini-Sling Versus Standard Midurethral Slings for Female Stress Urinary Incontinence: A Systematic Review and Meta-Analysis. Int Neurourol J. 2015 Dec;19(4):246-58. doi: 10.5213/inj.2015.19.4.246. Epub 2015 Dec 28. PMID 26739179
- [Background] Ellington DR, Erekson EA, Richter HE. Outcomes of Surgery for Stress Urinary Incontinence in the Older Woman. Clin Geriatr Med. 2015 Nov;31(4):487-505. doi: 10.1016/j.cger.2015.06.006. Epub 2015 Jul 26. PMID 26476111
- [Background] Jones KA, Harmanli O. Pessary use in pelvic organ prolapse and urinary incontinence. Rev Obstet Gynecol. 2010 Winter;3(1):3-9. PMID 20508777
- [Background] Bradley CS, Rahn DD, Nygaard IE, Barber MD, Nager CW, Kenton KS, Siddiqui NY, Abel RB, Spino C, Richter HE. The questionnaire for urinary incontinence diagnosis (QUID): validity and responsiveness to change in women undergoing non-surgical therapies for treatment of stress predominant urinary incontinence. Neurourol Urodyn. 2010 Jun;29(5):727-34. doi: 10.1002/nau.20818. PMID 19787711
- [Background] Hahn I, Fall M. Objective Quantification of Stress Urinary Incontinence: A Short Reproducible, Provocative Pad-Test. Neurourology and urodynamics. 1991;10:475-81.

RESULTS

PARTICIPANT FLOW:
Groups:
- With Yoni.Fit First: Yoni.Fit first, then without the Yoni.Fit.
- Without Yoni.Fit First: Without Yoni.Fit first, then with Yoni.Fit.
Period: Initial Assignment
Arm/Group | With Yoni.Fit First | Without Yoni.Fit First
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Cross Over
Arm/Group | With Yoni.Fit First | Without Yoni.Fit First
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- With Yoni.Fit First: With the Yoni.Fit first, then without the Yoni.Fit.
- Without Yoni.Fit First: Without the Yoni.Fit first, then with the Yoni.Fit.
- Total: Total of all reporting groups
Arm/Group | With Yoni.Fit First | Without Yoni.Fit First | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pad Weight Difference
Description: Comparison of urine weight of the pad without Yoni,Fit to the weight of the pad with Yoni.Fit controlling for the tare weight.
Time Frame: An hour after finishing a liter of liquid
Measure: Number; unit: grams
Groups:
- With Yoni.Fit: Pad weights for with the Yoni.Fit
- Without Yoni.Fit: Pad weights without Yoni.Fit.
Arm/Group | With Yoni.Fit | Without Yoni.Fit
Number analyzed (Participants) | 8 | 8
grams
  Subject #1 | 0.0 | 0.0
  Subject #2 | 0.0 | 0.3
  Subject #3 | 0.1 | 2.4
  Subject #4 | 0.3 | 0.4
  Subject #5 | 0.1 | 10.5
  Subject #6 | 0.1 | 6.0
  Subject #7 | 0.2 | 0.0
  Subject #8 | 17.3 | 9.2
Statistical Analysis 1: Comparison: With Yoni.Fit vs Without Yoni.Fit; Null hypothesis is that the pad weights With Yoni.Fit and Without Yoni.Fit are equivalent. A one-sided Wilcoxson paired T-test of the group means will be performed. If the p-value is significant, the null hypothesis will be rejected; Test type: Superiority; p = 0.0469, Wilcoxon (Mann-Whitney) — One subject experienced incontinence with the Yoni.Fit in place (#8) (9.2 g Pad Wt. Without and 17.3 g Pad Wt. With). This was attributed to incorrect Yoni.Fit sizing. This subject was not included in the p-value calculation

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- With Yoni.Fit: Those subjects assigned to use the Yoni.Fit first
- Without Yoni.Fit: Those subjects assigned to use the pad first.
Arm/Group | With Yoni.Fit | Without Yoni.Fit
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT03010800/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT03010800/ICF_001.pdf